CLINICAL TRIAL: NCT02435875
Title: The Analysis of Perioperative Baroreflex Sensitivity in Hypertensives
Brief Title: Perioperative Baroreflex Sensitivity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, DAN HUANG, Dr., RenJi Hospital
Other Study IDs: Renji1501
Record Dates: First submitted 2015-04-15; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension; Hemodynamic Instability; Surgery
Keywords: hypertension; perioperative; baroreflex sensitivity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hypertensive: Patients with confirmed hypertension or systolic blood pressure≥140 mmHg or diastolic blood pressure≥90 mmHg without antihypertensive treatment.After anesthesia induction,baroreflex sensitivity will be measured by nitroglycerin.
  Interventions: Other: no intervention
- nonhypertensive: systolic blood pressure <140 mmHg and diastolic blood pressure<90 mmHg.After anesthesia induction,baroreflex sensitivity will be measured by nitroglycerin.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Antihypertensive drug as intervention is used to see if it can improve baroreflex sensitivity to stable perioperative hemodynamic

SUMMARY:
Impaired baroreflex sensitivity (BRS) is a marker of autonomous dysfunction, which may play an important role in the long-term development of hypertension. Perioperative patients with hypertension is rapidly growing in all populations worldwide. However, no study has reported the values of BRS in this cohort. The aim of this study was to estimate the value of BRS for hypertension in a surgery cohort.

DETAILED DESCRIPTION:
Hypertension is known to be a major risk factor of end-organ damage, stroke and coronary mortality.It is estimated that one in six people worldwide, or nearly one billion, are affected by high blood pressure, and it is estimated that this number will increase to 1.5 billion by 2025. The World Health Organization also stated that high blood pressure is the most attributable cause of cardiovascular death.As the speed of aging is accelerated, the amount of perioperative hypertensive patients continue to increase. Perioperative hypertension had been shown to be a risk factor for the development of perioperative morbidity and mortality.Although it has aroused people's attention, there still lack of system evaluation and effective control. Therefore, it's urgent and necessary to assess and intervene perioperative situation of hypertensive patients.

The pathogenesis of hypertension is very complex, while the exact mechanism is still unclear. The dysfunction of autonomic activity, marked in particular by sympathetic overactivity and reduced parasympathetic activity, has been hypothesized to underlie the development of hypertension.Baroreflex control is one of the key mechanisms responsible for the short-term control of blood pressure.It acts as a closed loop, negative feedback mechanism, aimed at stabilizing blood pressure around a set point value.The impairment of baroreflex sensitivity (BRS) is know as the predictive factor of mortality in hypertension. A large of clinical and basic research indicated the existence of autonomic dysfunction and impaired BRS in patients with essential hypertension.

However, no study has reported the values of perioperative BRS, especially in hypertensive patients . Therefore, the aim of this study was to estimate the value of BRS for hypertension in a surgery cohort, and to explore the functional status of autonomic nervous system, may provide reference for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing ordinary thoracic surgery and age between 18 and 70;
2. American society of anesthesiologists(ASA) classification I to II level;
3. Willing to participate in this study and signed an informed consent

Exclusion Criteria:

1.Patients with diabetes mellitus, cardiopulmonary dysfunction, severe liver and kidney dysfunction and disease of nervous system;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing ordinary thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
baroreflex sensitivity | during operation
  Baroreflex sensitivity will be measured at three points include preoperation,intraoperation and postoperation

SECONDARY OUTCOMES:
interoperation complication | during operation
  Assessment of the incident of severe arrhythmia and blood pressure fluctuations
length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 5 days
  This assess how long patients stay in hospital
post-operative complications | 3 days postoperation
  Assessment of the incident of myocardial infarction,cerebral infarction and renal failure
hospitalization costs | 2 weeks postoperation
  Hospitalization costs will be assessed after patients discharged from hospital

CONTACTS AND LOCATIONS:
Overall Officials: WEIFENG YU, MD, Study Chair — Anesthesiology Department Renji Hospital, Shanghai Jiao Tong University, School of Medicine
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China